CLINICAL TRIAL: NCT00761995
Title: Safety and Efficacy of Brinzolamide Dosed TID With Dorzolamide Dosed TID in Reducing Intraocular Pressure in Patients With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-CT-08-003
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-01

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Raised IOP
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — brinzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azopt (Active Comparator): topical eye drop dosed 1 drop 3 times daily
  Interventions: Drug: Azopt
- Cosopt (Active Comparator): topical eye drop
  Interventions: Drug: Cosopt

INTERVENTIONS:
Drug: Azopt — topical eye drop dosed 1 drop 3 times daily
  Arms: Azopt
Drug: Cosopt — topical eye drop dosed 1 drop 2 times daily
  Arms: Cosopt

SUMMARY:
Safety and Efficacy of Brinzolamide Dosed TID With Dorzolamide Dosed TID in Reducing Intraocular Pressure in Patients With Open Angle Glaucoma or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years of age or older, diagnosed with primary open-angle glaucoma or ocular hypertension.
* If of child bearing potential

  * Must use a reliable means of contraception for the duration of the study or surgically sterilized.
* Must have a negative pregnancy test.
* Must be non-lactating
* IOP measurements ≥ 24 ≤ 36 mm Hg, in at least one eye, at 9.00 a.m and ≥ 21 ≤ 36 mm Hg in at least one eye (the same eye) at 11.00 am measurement
* The IOP criteria to be met at both time points by the same eye
* Visual Acuity of 6/24 or better in study eye (s)
* Gonioscopy angle of ≥ 2 in the study eye (s)
* Patients with a level of understanding and willingness to fully comply with all visits and study procedures scheduled by the study site as evidenced by written informed consent

Exclusion Criteria:

* Patients with one sighted eye or amblyopia
* History of chronic or recurrent uveitis or other inflammatory eye disease (e.g. scleritis).
* History of ocular infections (e.g. conjunctivitis) within past 3 months.
* History of ocular trauma within the past 6 months.
* History of severe or progressive retinal (i.e. retinal degeneration, diabetic retinopathy, retinal detachment or retinal tears) or optic nerve disease.
* History of severe ocular pathology such as severe glaucoma damage determined by optic nerve head (e.g. C/D ratio > 0.8) or visual field evaluation (e.g. split fixation, clinically significant field loss within the central field) or legal blindness in either eye.
* Intraocular surgery within the past 12 months or Laser surgery within the past 3 months as determined by patient history and/or examination.
* Any other form of glaucoma other than primary open angle glaucoma.
* Inability to discontinue contact lens wear during the day
* History of hypersensitivity to oral or topical CAIs, sulfonamide drugs or to any component of these medicines.
* Any abnormality preventing reliable applanation tonometry of either eye.
* Patients who are in the investigator's best judgement at risk of visual field or visual acuity worsening as a consequence of participation of trial.
* Chronic use of any systemic medication that may effect IOP with less than one month stable dosing regimen (i.e. sympathomimetic agents, beta-adrenergic blocking agents, alpha agonists, alpha-adrenergic blocking agents, calcium channel blockers, angiotensin-converting enzyme inhibitors, etc.).
* Current use of any ophthalmic, dermatologic or systemic steroid.
* Patients with clinically significant medical (acute or progressive) condition e.g. cardiovascular, pulmonary, hematologic disease or psychiatric illness, who are unlikely to fully complete all protocol requirements as assessed by the investigator.
* Participation in another clinical trial within past 30 days.
* Pregnant and lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
IOP reduction from baseline at the end of 12 weeks | 12 weeks

SECONDARY OUTCOMES:
IOP reduction from baseline at the end of 4 and 8 weeks of treatment | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Laboratories, India, Bangalore, India